CLINICAL TRIAL: NCT04152161
Title: A Randomized, Placebo Controlled, Observer-Blind, Phase IIb Study to Evaluate the Efficacy, Safety, and Immunogenicity of BCG Revaccination in Healthy Adolescents for the Prevention of Sustained Infection With Mycobacterium Tuberculosis
Brief Title: Bacille Calmette Guerin (BCG) Revaccination of Healthy Adolescents for the Prevention of Mycobacterium Tuberculosis Sustained Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gates MRI-TBV01-201
Record Dates: First submitted 2019-10-22; First posted 2019-11-05 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis infection; Healthy adolescents; Healthy participants; BCG vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bacille Calmette Guerin (BCG) group (Experimental)
  Interventions: Biological: BCG vaccine SSI
- Placebo group (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BCG vaccine SSI — Participants will receive a single 0.1 milliliter (mL) volume of BCG vaccine SSI, administered intradermally in deltoid region of the upper arm.
  Arms: Bacille Calmette Guerin (BCG) group
Biological: Placebo — Participants will receive a single 0.1 mL volume of normal saline, administered intradermally in deltoid region of the upper arm.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to demonstrate the efficacy of Bacille Calmette Guerin (BCG) revaccination against sustained Mycobacterium tuberculosis infection versus placebo in previously BCG vaccinated QuantiFERON®-TB Gold Plus Assay (QFT) negative, healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Participant between ≥ 10 years and ≤ 18 years on Study Day 1
* General good health, confirmed by medical history and physical examination
* Vaccinated with Bacille Calmette Guerin (BCG) at least 5 years ago, documented through medical history or by presence of healed BCG scar
* Tests QuantiFERON®-TB Gold Plus Assay (QFT) negative at screening.
* For female participants: not pregnant and agrees to avoid pregnancy throughout the first 12 months of the study. Women physically capable of pregnancy must agree to use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include sexual abstinence (not engaging in sexual intercourse), a confirmed sterile partner, or at least 2 contraception methods from the following list: male or female condom, diaphragm, intrauterine devices (IUDs), hormonal contraceptive (oral, injection, transdermal patch, or implant).
* Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
* Capable of giving signed informed consent/assent and completes the written informed consent/assent process.

Exclusion Criteria:

* Acute illness on Study Day 1. NOTE: This is a temporary exclusion for which the participant may be re-evaluated
* Body temperature ≥37.5 degree Celsius on Study Day 1. NOTE: This is a temporary exclusion for which the participant may be re-evaluated
* History or evidence of any clinically significant disease, including severe eczema and severe asthma, or any acute or chronic illness that might affect the safety, immunogenicity, or efficacy of study vaccine in the opinion of the investigator
* Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol
* History of autoimmune disease
* History or evidence of active tuberculosis (TB) disease
* History or laboratory evidence of any past or present possible immunodeficiency state including, but not limited to, any laboratory indication of human immunodeficiency virus - 1 (HIV-1) infection
* History of allergic disease that is likely to be exacerbated by any component of the study vaccine
* History of treatment for active TB disease or history of latent Mycobacterium tuberculosis infection
* Received a tuberculin skin test within 6 months prior to Study Day 1
* Received immunosuppressive treatment, e.g., chemotherapy, biologics or radiation therapy, or used immunosuppressive medication (daily steroid equivalent of ≥5 milligrams prednisone) within 42 days before Study Day 1. Inhaled and topical corticosteroids are permitted.
* Received immunoglobulin or blood products within 42 days before Study Day 1
* Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 28 days after Study Day 1
* Received investigational TB vaccine at any time prior to Study Day 1
* Received any investigational drug therapy or investigational vaccine within 180 days before Study Day 1, or planned participation in any other clinical trial using investigational product during the study period
* Laboratory values from the most recent blood collected prior to randomization outside the normal range that are suggestive of a disease state. Grade 1 abnormalities (as per Division of Acquired Immunodeficiency Syndrome toxicity table version 2.1) do not lead to exclusion if the investigator considers them not clinically significant
* Urinalysis abnormality greater than Grade 1 on the Toxicity Scale (with the exception of hematuria in a menstruating female), or urinalysis abnormality judged clinically significant by the investigator
* Shared residence with an individual who is receiving TB treatment or with someone who is known to have incompletely treated TB. e.g., Xpert Mycobacterium tuberculosis (MTB)/rifampicin (RIF) assay-positive, polymerase chain reaction-positive, culture-positive, smear-positive TB, or clinically diagnosed unconfirmed TB
* Child in Care
* Female participants currently pregnant or lactating/nursing; or positive serum pregnancy test during screening or on Day 1, prior to vaccination, or planning a pregnancy within the first 12 months after study intervention

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1836 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (5):
- South Africa (5):
  - Investigational Site, Klipfontein, Cape Town
  - Investigational Site, Berea, Durban
  - Investigational Site, Hillbrow, Johannesburg
  - Investigational Site, Paarl, Western Cape
  - Investigational Site, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Schmidt AC, Fairlie L, Hellstrom E, Luabeya Kany Kany A, Middelkoop K, Naidoo K, Nair G, Gela A, Nemes E, Scriba TJ, Cinar A, Frahm N, Mogg R, Kaufman D, Dunne MW, Hatherill M; BCG REVAX Study Team. BCG Revaccination for the Prevention of Mycobacterium tuberculosis Infection. N Engl J Med. 2025 May 8;392(18):1789-1800. doi: 10.1056/NEJMoa2412381. PMID 40334156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIb, randomized, placebo-controlled, observer-blind study to evaluate the efficacy, safety, and immunogenicity of Bacille Calmette Guerin (BCG) revaccination against sustained Mycobacterium tuberculosis infection versus placebo in previously BCG vaccinated QuantiFERON®-TB Gold Plus Assay (QFT) negative, healthy adolescents.
Pre-assignment Details: A total of 1836 participants were enrolled from South African and were randomized 1:1 to experimental and placebo groups.
Groups:
- Bacille Calmette Guerin (BCG) Group: Participants were randomized to receive a single 0.1 milliliter (mL) volume of BCG vaccine Statens Serum Institut (SSI), administered intradermally in deltoid region of the upper arm.
- Placebo Group: Participants were randomized to receive a single 0.1 mL volume of normal saline, administered intradermally in deltoid region of the upper arm.
Period: Overall Study
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Started | 919 | 917
Did Not Receive the Intervention | 1 | 0
Completed | 110 | 111
Not Completed | 809 | 806
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 9 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 29 | 28
Not completed — Sponsor termination of study | 750 | 755
Not completed — Other | 20 | 18

BASELINE CHARACTERISTICS:
Population: Safety Population comprises of all participants who received the study intervention.
Groups:
- Bacille Calmette Guerin (BCG) Group: Participants were randomized to receive a single 0.1 mL volume of BCG vaccine SSI, administered intradermally in deltoid region of the upper arm.
- Total: Total of all reporting groups
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group | Total
Number analyzed (Participants) | 918 | 917 | 1835
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.4 (1.68) | 13.4 (1.67) | 13.4 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 474 | 469 | 943
  Male | 444 | 448 | 892
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 625 | 627 | 1252
  Unknown or Not Reported | 292 | 290 | 582
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 729 | 735 | 1464
  Asian Indian | 0 | 1 | 1
  Mixed Race | 63 | 61 | 124
  Southern African Colored | 125 | 120 | 245
  White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained QuantiFERON®-TB Gold Plus Assay (QFT) Conversion From a Negative to Positive Test Based on Positive QFT Test Results
Description: Sustained conversion was defined as sustained QFT conversion from a negative to positive test, with initial conversion at any time after a first negative QFT result post randomization (Day 71 or subsequent visit if Day 71 result was not available), and remaining QFT positive at 3- and 6-months post-conversion.
Time Frame: Up to 48 months
Population: Modified Intention to Treat Efficacy Population comprised of all participants randomly assigned to study intervention who received the study intervention, and are QFT negative at the Day 71 visit, or at the first study visit post Day 71 for which a QFT result is available if the Day 71 study visit was missed or the Day 71 QFT result was not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 871 | 849
Participants | 82 | 78
Statistical Analysis 1: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; Vaccine Efficacy = -0.049, 95% CI 2-sided [-0.431 to 0.230] — Vaccine Efficacy (VE) = 1 - Hazard Ratio, with 95%CI equal to (VE lower limit, VE upper limit) = (1 - Hazard Ratio upper limit, 1 - Hazard Ratio lower limit)
Statistical Analysis 2: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; p = 0.6193, Log Rank; The 1-sided p-value from the log-rank test was stratified by sex and age group; Hazard Ratio (HR) = 1.049, 95% CI 2-sided [0.770 to 1.431] — Hazard ratio was calculated using a stratified Cox proportional hazards model, with sex and age group (10-11 years, 12-14 years, and >14 years) as stratification variables

2. Secondary Outcome: Number of Participants With Sustained QFT Conversion From a Negative to Positive Test Based on Positive QFT Test Results at 36-Months Follow-up or Discontinued Early
Description: as for outcome 1
Time Frame: 36 Months Follow-up
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 871 | 849
Participants | 74 | 73
Statistical Analysis 1: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; Vaccine Efficacy = -0.009, 95% CI 2-sided [-0.395 to 0.270] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; p = 0.5224, Log Rank; The 1-sided p-value from the log-rank test was stratified by sex and age group; Hazard Ratio (HR) = 1.009, 95% CI 2-sided [0.730 to 1.395] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Number of Participants With Sustained QFT Conversion From a Negative to Positive Test Based on Positive QFT Test Results at 48-Months Follow-up or Discontinued Early
Description: as for outcome 1
Time Frame: 48 Months Follow-up
Population: mITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Bacille Calmette Guerin (BCG) Group: Participants were randomized to receive a single 0.1 milliliter (mL) volume of BCG vaccine SSI, administered intradermally in deltoid region of the upper arm.
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 871 | 849
Participants | 82 | 78
Statistical Analysis 1: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; Vaccine Efficacy = -0.049, 95% CI 2-sided [-0.431 to 0.230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bacille Calmette Guerin (BCG) Group vs Placebo Group; Test type: Superiority; p = 0.6193, Log Rank; The 1-sided p-value from the log-rank test was stratified by sex and age group; Hazard Ratio (HR) = 1.049, 95% CI 2-sided [0.770 to 1.431] — Calculated using a stratified Cox proportional hazards model, with sex and age group (10-11 years, 12-14 years, and >14 years) as stratification variables

4. Secondary Outcome: Number of Participants With Serious and Non-serious Solicited Adverse Events (AEs) Through 7 Days Post Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE does not necessarily have a causal relationship with the intervention. Solicited AEs were defined as events that participants were specifically asked about and which were noted by participants in the diary card. Solicited AEs included injection site symptoms of injections site pain, redness and swelling and general body symptoms such as headache, fatigue, gastrointestinal symptoms, and fever.
Time Frame: Day 1 through Day 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 918 | 917
Participants
  Any injection site symptom | 754 | 381
  Any general body symptom | 371 | 314

5. Secondary Outcome: Number of Participants With Unsolicited AEs Through Day 28, as Well as Solicited AEs That Were Ongoing at Day 7 After Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE does not necessarily have a causal relationship with the intervention. Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary card, as well as solicited AEs that were ongoing at Day 7 after vaccination. Number of Participants With Unsolicited AEs Through 28 Days after vaccination has been presented.
Time Frame: Day 1 through Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 918 | 917
Participants | 185 | 117

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of Participants reporting SAEs has been presented.
Time Frame: Up to 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 918 | 917
Participants | 3 | 3

7. Secondary Outcome: Number of Participants With AEs of Special Interest
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AE of special interest are AEs that the sponsor closely monitors. The AEs of special interest to be collected and reported include immune system disorders (anaphylactic reaction), general disorders (disseminated BCG disease), infections and infestations (osteomyelitis, suppurative lymphadenitis, injection site abscess), skin and subcutaneous tissue disorders (injection site lupus vulgaris, injection site keloid formation), and bone disorders (osteitis).
Time Frame: Up to 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 918 | 917
Participants
  Injection site abscess | 4 | 0
  Suppurative lymphadenitis (Lymphadenitis bacterial) | 1 | 0
  Anaphylactic reaction | 0 | 0
  Disseminated BCG disease | 0 | 0
  Osteomyelitis | 0 | 0
  Injection site lupus vulgaris | 0 | 0
  Injection site keloid formation | 0 | 0
  Osteitis | 0 | 0

8. Secondary Outcome: Number of Participants With Serious Adverse Drug Reactions (ADRs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. When an AE is judged to be serious and related to an investigational product, it is a Serious ADR.
Time Frame: Up to 48 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
Number analyzed (Participants) | 918 | 917
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs (comprising of injection site pain, redness, swelling, headache, fatigue, gastrointestinal symptoms, and fever) were recorded on diary cards (systematic assessment) for 7 days after vaccination. Solicited events ongoing at Day 7 were also recorded as unsolicited AEs. Unsolicited AEs were collected through Day 28, SAEs and All-cause mortality through Month 6 and Serious adverse drug reactions (ADRs) through Month 48.
Description: Serious adverse events and non-serious adverse events were collected in Safety Population. An AE was classified as solicited if it was proactively recorded through a structured assessment (e.g., diary card) through 7 days post vaccination. Unsolicited AEs collected outside the daily card were presented separately. A participant who had a solicited event that was ongoing at Day 7 would have the event counted as both a solicited AE and an unsolicited AE.
Arm/Group | Bacille Calmette Guerin (BCG) Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/918 | 1/917
Serious Adverse Events (participants affected / at risk) | 3/918 | 3/917
Other Adverse Events (participants affected / at risk) | 800/918 | 540/917
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bacille Calmette Guerin (BCG) Group (N=918) | Placebo Group (N=917)
Sinusitis (Infections and infestations) | 1 | 0
Subperiosteal abscess (Infections and infestations) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bacille Calmette Guerin (BCG) Group (N=918) | Placebo Group (N=917)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 136 | 140
Injection site swelling (General disorders) | 657 | 248
Injection site pain (General disorders) | 381 | 148
Injection site erythema (General disorders) | 349 | 111
Fatigue (General disorders) | 229 | 184
Injection site ulcer (General disorders) | 20 | 0
Pyrexia (General disorders) | 24 | 27
Injection site pain (General disorders) | 21 | 0
Pyrexia (General disorders) | 12 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 15
Headache (Nervous system disorders) | 195 | 164
Headache (Nervous system disorders) | 36 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT04152161/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT04152161/SAP_001.pdf